CLINICAL TRIAL: NCT06727097
Title: Tracking the Development and Influence of Post-Stroke Sensory Reweighting on Walking and Balance Outcomes
Brief Title: Post-Stroke Sensory Reweighting on Walking and Balance Outcomes
Acronym: PSR
Status: Recruiting | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Oluwole Awosika, Principal Investigator, University of Cincinnati
Other Study IDs: 2024-0585; 1R21HD115776-01 (NIH)
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Walking Speed; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Stroke Survivors: First ever clinical stroke (ischemic, supratentorial, and unilateral)
  Interventions: Diagnostic Test: Posturography; Diagnostic Test: Walking Speed; Diagnostic Test: Instrumented 7M Timed UP and GO; Other: Fall Event Records; Diagnostic Test: MRI (3T)

INTERVENTIONS:
Diagnostic Test: Posturography — Successful completion of all four indices of the mCTSIB, without severe imbalance (i.e., near fall with safety harness and urgent knee to grab emergency handlebars) constitutes "PSR +", non-completing on any of the index is noted as "PSR -". Exploratorily, the average sway velocity index will be captured for each condition, to characterize sensory reweighting patterns.
  Other Names: mCITSIB
Diagnostic Test: Walking Speed — The 10-meter walk test (10MWT) is the gold standard measure of post-stroke walking function that reflects overall mobility and health status. Method: Two 10MWT trials (using a stopwatch) are averaged and documented in meters/second. The functional ambulatory category (FAC) will be collected as supplement. Exploratorily: Participants will also perform the 10mWT (fast paced-FP) with two attempts. Both SS and FP will be performed over the Zeno Walkway Gait Analysis Mat, to capture supplementary spatiotemporal data.
  Other Names: 10 Meter Walk Test
Diagnostic Test: Instrumented 7M Timed UP and GO — This sub-aim will use iTUG to determine the effects of BLT on dynamic balance. In contrast to the traditional TUG, inclusion of wearable triaxial accelerometers and gyroscopes-placement test increases the sensitivity (87%) and specificity (87%) for identifying individuals prone to falls. Two trials are averaged and documented in seconds. Secondary analysis will be performed on data obtained from the sensors to determine (stride length, stride velocity, cadence, peak arm swing velocity, and turning velocity, during the task), to correlate with the TUG time/speed. Time points: Same as Posturography and 10 MWT.
  Other Names: iTUG
Other: Fall Event Records — A robust fall incident journal elucidating the date, time, nature, and management of the fall event will be provided to all study participants for documentation. The study research coordinator will contact the patient/caregiver/facility to collect the data q2 weeks. A tally of the total number of fall events between visits will be recorded.
Diagnostic Test: MRI (3T) — Structural neuroimaging biomarkers:. The fractional anisotropy map from the primary fiber population in each voxel will be resampled to MNI space (using the warp derived from structural preprocessing) and projected onto a template white matter skeleton using local maxima to further optimize registration accuracy. Small vessel disease parameters, including white matter hyperintensities using the Fazekas scale and number/site of microhemorrhages, will be recorded for exploratory analyses.

SUMMARY:
The primary objective of this proof-of-concept study is to longitudinally track the development of post-stroke sensory reweighting (PSR), identify associated structural neuroanatomical correlates, and investigate their relationship to walking and fall outcomes.

DETAILED DESCRIPTION:
Post-stroke imbalance and walking impairment is a function of diminished sensorimotor integration, motor, and postural control. It impacts over 75% of stroke survivors, and remain a rising cause of falls, fractures, and death in the United States. The associated fear of falling often leads to a downward spiral of health, characterized by reduced walking performance, caregiver dependency, social isolation, and the development of secondary post-stroke medical complications. Although spontaneous biological recovery and intensive clinical rehabilitation may improve balance and walking ability, the extent of recovery is often limited after the first 6-months of stroke (chronic phase). Furthermore, currently available clinical measures such as the Berg Balance Scale and Timed-Up-and-Go lack the specificity and granularity needed to foster the development of individualized and targeted neurorehabilitation interventions. In addition, non-invasive neurostimulation strategies lack specificity due to limited understanding of the most appropriate neuroanatomical targets for optimizing sensorimotor integration. Hence there is an urgent need to identify reliable physiologic and neuroanatomic correlates in the earlier stages of recovery (<6 months), to enable timely and targeted rehabilitation interventions.

ELIGIBILITY:
Inclusion Criteria:

1. First ever clinical stroke
2. Stroke due to ischemia
3. Age 18 years or older
4. Ability to consent by patient (not surrogate), any time prior to acute hospital discharge

Exclusion Criteria:

1. Pre-stroke dependence (modified Rankin Scale score of 3 or more)
2. Isolated brainstem or cerebellar stroke
3. Bilateral acute strokes
4. Co-enrollment in a trial of an intervention through six-month follow-up
5. Inability to maintain follow-up with study procedures through six-month follow-up
6. Contraindication to non-contrast MRI
7. Low likelihood of survival beyond the acute hospitalization, such as malignant cerebral edema
8. Pre-existing co-morbid conditions that significantly affects vision, somatosensory function, vestibular system, orthostasis, coordination or mobility
9. Post stroke mRS>4 or discharge to hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic Stroke (unilateral, Supratentorial)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Posturography | 2, 4, and 6 months Post-Stroke
  MCTSIB
Walking Speed (10 meter Walk Test) | 2, 4, and 6 months Post-Stroke
  Self-Selected
Instrumented Timed UP and GO | 2, 4, and 6 months Post-Stroke
  7M ITUG
Fall Events | 2, 4, and 6 months Post-Stroke
  Record and characterization of Falls

SECONDARY OUTCOMES:
Functional Ambulation Category | 2, 4, and 6 months Post-Stroke
  Determination of walking status
Walking Speed (10 meter Walk Test) | Walking Speed (10 meter Walk Test)
  Fastest Speed

CONTACTS AND LOCATIONS:
Overall Officials: Oluwole Awosika, MD, MSCR, Principal Investigator — University of
Locations (1):
- University of Cincinnati College of Medicine, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No